CLINICAL TRIAL: NCT07078695
Title: A Phase 1, Randomized, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single Subcutaneous/Intravenous Administered SHR-1139 in Healthy Participants
Brief Title: A Trial of SHR-1139 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1139-102
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1139 dose level 1 (Experimental): Single dose of SHR-1139 given subcutaneously (dose level 1)
  Interventions: Drug: SHR-1139 Injection
- SHR-1139 dose level 2 (Experimental): Single dose of SHR-1139 given subcutaneously (dose level 2)
  Interventions: Drug: SHR-1139 Injection
- SHR-1139 dose level 3 (Experimental): Single dose of SHR-1139 given intravenously (dose level 3)
  Interventions: Drug: SHR-1139 Injection

INTERVENTIONS:
Drug: SHR-1139 Injection — Single dose of SHR-1139 given subcutaneously (dose level 1 )
  Arms: SHR-1139 dose level 1
Drug: SHR-1139 Injection — Single dose of SHR-1139 given subcutaneously (dose level 2 )
  Arms: SHR-1139 dose level 2
Drug: SHR-1139 Injection — Single dose of SHR-1139 given intravenously (dose level 3)
  Arms: SHR-1139 dose level 3

SUMMARY:
The purpose of this study is to assess safety, PK and immunogenicity profile of a single dose of SHR-1139 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy white participants.
2. Ability to understand the trial procedures and possible adverse events, volunteer to participate in the trial, and provide written informed consent, be able to comply with all the requirements, and able to complete the study.
3. Male aged between 18 to 55 years of age (inclusive)
4. Women with body weight ≥ 45.0 kg, men with body weight ≥ 50.0 kg, body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening.
5. Men and WOCBP must agree to take highly effective contraceptive methods

Exclusion Criteria:

1. History or evidence of clinically significant disorders.
2. Individuals with a history of drug allergies, specific allergies, or known history or suspected of being allergic to the study drug or any component of it.
3. Receipt of medical devices or another investigational drug (including placebo) within 3 months or 5 half-lives, or in the follow-up period of a clinical study, whichever is longer (according to the date of the signed consent form) prior to screening.
4. Unwilling or unable to comply with the Lifestyle Guidelines detailed in this protocol.
5. Positive pregnancy test at screening or D-1/check-in.
6. Any other circumstances (e.g., not suitable for venous access) or laboratory abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PK profile of SHR-1139 after a single administration | Start of Treatment to end of study (Day 253)
  Pharmacokinetics- Area under the concentration-time curve from time 0 to last time point after SHR-1139 administration (AUC0-last)
PK profile of SHR-1139 after a single administration | From time 0 to infinity after SHR-1139 administration (Day 253)
  Pharmacokinetics- Area under the concentration-time curve (AUC0-inf)
PK profile of SHR-1139 after a single administration: | Start of Treatment to end of study (Day 253)
  Pharmacokinetics- Time to Cmax of SHR-1139 (Tmax )
PK profile of SHR-1139 after a single administration | Start of Treatment to end of study (Day 253)
  Pharmacokinetics-Terminal elimination half-life of SHR-1139 (t1/2)
Immunogenicity profile of SHR-1139 after a single dose administration | Day 253
  The number of participants with anti-drug antibody (ADA)

SECONDARY OUTCOMES:
Safety and Tolerability Based on Incidence and Severity of Treatment Emergent Adverse Events | Day 295
  Number of participants with Adverse events and Serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Linear, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No